CLINICAL TRIAL: NCT04987112
Title: A Phase 1, Dose Escalation, Open-Label Study of Intratumoral CAN1012 in Subjects With Unresectable or Metastatic Advanced Solid Tumors
Brief Title: Intratumoral CAN1012(Selective TLR7 Agonist) in Subjects With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CanWell Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN1012
Record Dates: First submitted 2021-07-09; First posted 2021-08-03 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Solid Tumor; Cancer Metastatic
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAN1012 single agent (Experimental): CAN1012 intratumoral injection given alone
  Interventions: Drug: CAN1012

INTERVENTIONS:
Drug: CAN1012 — CAN1012 IT injection (once every 4 weeks)

SUMMARY:
To evaluate CAN1012(Selective TLR7 agonist) when administered by IT injection to subjects with advanced solid tumors who are not candidates for standard therapy.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, first-in-human, single-arm, multicenter, dose escalation study of IT CAN1012 in subjects with advanced solid tumors who are not candidates for standard therapy.

Subjects will be enrolled in cohorts of 3 at each dose level using a 3+3 dose escalation design Approach.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and willing to comply with the study's requirements.
2. Male or female age >18 years at screening.
3. Metastatic or locally advanced solid tumor that has progressed on, is refractory to, or for which there is no efficacious standard of care therapy.
4. Demonstrate adequate organ function as defined below. All screening laboratory assessments should be performed within 14 days of treatment initiation.
5. Performance status of 0 or 1 on the ECOG Performance Scale.
6. Life expectancy >12 weeks at Baseline.
7. Women of childbearing potential must have negative serum pregnancy test within 3 days prior to receiving the first study drug administration.
8. For women of childbearing potential, must be willing to use an adequate method of contraception from 30 days prior to the first study drug administration and 120 days following last day of study drug administration.
9. Male subjects of childbearing potential must be surgically sterile or must agree to use adequate method of contraception during the study and at least 120 days following the last day of study drug administration.

Exclusion Criteria:

1. Received prior TLR7/8 agonists (excluding topical agents).
2. Has untreated or uncontrolled central nervous system (CNS) involvement.
3. Will receive concurrent chemotherapy, immunotherapy, biologic, hormonal therapy, or other therapies for cancer.
4. Received systemic interferon alfa (IFNα) prior to enrollment.
5. Unresolved toxicities from prior therapy, defined as having not resolved to CTCAE v5.0 Grade 0 or 1, with exception of endocrinopathies from prior therapy, alopecia, and vitiligo.
6. Treatment with systemic corticosteroids.
7. Concomitant or planned use of sensitive substrates of major cytochrome P450 enzymes.
8. Has an active infection requiring systemic therapy.
9. Has known active infection with the human immunodeficiency virus,
10. Unstable/inadequate cardiac function.
11. Uncontrolled concurrent illness.
12. A history of interstitial lung disease.
13. A history of coagulopathy resulting in uncontrolled bleeding or other bleeding disorders.
14. Participated in a clinical study of an investigational agent within 30 days of screening.
15. Has known psychiatric, substance abuse, or other disorders that would interfere with cooperation with the requirements of the study in the opinion of the investigator.
16. Is pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 12 months
  Safety and tolerability as determined by assessment of dose limiting toxicities and the maximum tolerated dose or maximal assessed dose per protocol of CAN1012 with cancers.
Recommended Phase 2 Dose (RP2D) | 12 months
  To determine a recommended phase 2 dose of CAN1012 for further development by evaluating number of patients with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0)
Maximum Tolerated Dose (MTD) | 12 months
  Determine the maximum tolerated dose by assessing the Incidence of Dose Limiting Toxicities (DLTs), treatment emergent and treatment related adverse events (assessed by CTCAE v5.0).

SECONDARY OUTCOMES:
PK characterization - Cmax | 12 months
  Maximum observed plasma and tumor concentration of CAN1012 after IT administration.
PK characterization - tmax | 12 months
  Time to reach maximum plasma and tumor concentration of CAN1012 after IT administration.
tumor size in injected lesions and non-injected lesions | 12 months
  Changes in tumor size using computed tomography (CT) scan or magnetic resonance imaging (MRI) scan assessment based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - CanWellPharma, Woburn, Massachusetts
  - Providence Cancer Institute, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No